CLINICAL TRIAL: NCT03315208
Title: Pilot Study of a Transdiagnostic, Emotion-focused Group Intervention for Young Adults With Substance Use Disorders
Brief Title: Study of a Transdiagnostic, Emotion-focused Group Intervention for Young Adults With Substance Use Disorders
Acronym: ARMS UP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Kate Bentley, PhD, Assistant Professor, Harvard Medical School, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017P001274
Record Dates: First submitted 2017-10-04; First posted 2017-10-20 (Actual); Results first posted 2021-04-01 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Substance Use Disorders; Depression; Anxiety; Emotional Disorder; Suicidal Ideation; Suicidal and Self-injurious Behavior
Keywords: transdiagnostic treatment; cognitive-behavioral therapy; Unified Protocol; young adults; substance use disorder; emotional disorder; depression; anxiety; emotion dysregulation; self-injurious thoughts and behaviors
MeSH Terms: conditions — Substance-Related Disorders; Depression; Anxiety Disorders; Suicidal Ideation; Self-Injurious Behavior; Behavior | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Unified Protocol + Treatment As Usual (Experimental): Participants in this arm are offered 16 twice-weekly group UP sessions in addition to TAU at an existing comprehensive outpatient program for adolescents and young adults with substance use disorders.
  Interventions: Behavioral: Unified Protocol (UP); Other: Treatment as Usual (TAU)
- Treatment As Usual Alone (Active Comparator): Participants in this arm undergo TAU at an existing comprehensive outpatient program for adolescents and young adults with substance use disorders.
  Interventions: Other: Treatment as Usual (TAU)

INTERVENTIONS:
Behavioral: Unified Protocol (UP) — The Unified Protocol for Transdiagnostic Treatment of Emotional Disorders (UP) is an evidence-based psychological intervention designed to be applied across anxiety, depressive, and other disorders in which emotion dysregulation is central. The UP targets shared temperamental vulnerabilities to emotional disorders through emotion-focused CBT strategies.
  Arms: Unified Protocol + Treatment As Usual
Other: Treatment as Usual (TAU) — Treatment as Usual consists of some combination of group therapy, individual therapy, and/or psychopharmacology appointments at an existing comprehensive outpatient program for adolescents and young adults with substance use disorders.

SUMMARY:
The overall aim of this pilot study is to conduct a preliminary trial to evaluate the acceptability and feasibility of adding a transdiagnostic, emotion-focused group intervention (the Unified Protocol, UP) to treatment as usual (TAU) in a comprehensive outpatient program for adolescents and young adults with substance use disorders and emotional distress. Only patients seeking services or engaged in care at an existing outpatient program at MGH (the Addiction Recovery Management Service) are eligible for participation.

DETAILED DESCRIPTION:
Young adults with substance use disorder (SUD) commonly experience co-occurring emotional distress in the form of affective/emotional disorders (i.e. anxiety, depressive, and related disorders) and self-injurious thoughts and behaviors (SITBs). Based on the conceptualization of emotion dysregulation as a transdiagnostic treatment target, the current study utilizes the Unified Protocol for Transdiagnostic Treatment of Emotional Disorders (UP) to target core psychopathological processes related to emotion dysregulation that underlie SITBs and emotional disorder pathology. Given its transdiagnostic format, the UP has the potential to address comorbidity among the emotional disorders (and other functionally similar problems such as SUDs) simultaneously and more comprehensively than single-diagnosis treatments.

Patients seeking services or currently engaged in care at an existing comprehensive outpatient program for adolescents and young adults with substance use disorders (the MGH Addiction Recovery Management Service) are eligible for this study. Participants will be randomized 2:1 to receive either UP + TAU or TAU alone. The adjunctive UP intervention consists of 16 twice-weekly group sessions (delivered over an 8-week period) designed to deliver transdiagnostic, emotion-focused CBT strategies.

ELIGIBILITY:
Only patients seeking services or currently engaged in care at the MGH Addiction Recovery Management Service are eligible for this study.

Inclusion Criteria:

1. Young adults ages 18 to 26, inclusive
2. English language proficiency
3. Ability to provide written, informed consent
4. Ability to attend in-person, outpatient sessions
5. Has provided consent to receive or is currently undergoing treatment at the MGH Addiction Recovery Management Service
6. Documented DSM-5 SUD diagnosis (limited to alcohol use disorder; cannabis use disorder; phencyclidine or other hallucinogen use disorder; inhalant use disorder, opioid use disorder; sedative, hypnotic, or anxiolytic use disorder; stimulant use disorder; other (or unknown) SUD)
7. Current elevated emotional distress, as evidenced by any one of the following:

   1. Score at least in the moderate range on self-report anxiety questionnaire
   2. Score at least in the moderate range on self-report depression questionnaire
   3. Report of suicidal thoughts in the past week
   4. Report of engagement in non-suicidal self-injury in the past week
8. Not expected to require inpatient level of care within the next two weeks (as judged clinically)

Exclusion Criteria:

1. Documented psychotic disorder (or current, clinically significant psychotic symptoms) that render the patient inappropriate for outpatient level of care or participation in group therapy (as judged clinically by study staff)
2. Current imminent suicide or homicide risk (as judged clinically by study staff)
3. Unwilling or unable to provide consent for study staff to access subject's medical records and coordinate care and exchange data with clinical staff at the Addiction Recovery Management Service
4. Unwilling or unable to identify an emergency contact

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2017-11-22 (Actual); Primary Completion 2019-09-20 (Actual); Study Completion 2019-09-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eden Evins, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital Addiction Recovery Management Service, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from November 2017 to July 2019 from an outpatient treatment program for adolescents and young adults with substance use disorders.
Pre-assignment Details: Participants were randomized in cohorts of 5. Thus, participants underwent a "waiting to be randomized" period from enrollment until the date they were randomized.
  9 participants were excluded between the point of enrollment to randomization; 8 due to not meeting inclusion criteria, and 1 withdrawn by the PI while waiting to be randomized.
Period: Overall Study
Arm/Group | Unified Protocol + Treatment As Usual | Treatment As Usual Alone
Started | 29 | 18
Completed | 16 | 12
Not Completed | 13 | 6
Not completed — Lost to Follow-up | 11 | 6
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Unified Protocol + Treatment As Usual | Treatment As Usual Alone | Total
Number analyzed (Participants) | 29 | 18 | 47
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 29 | 18 | 47
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.6 (2.1) | 21.6 (1.9) | 21.6 (1.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 8 | 20
  Male | 17 | 10 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 1 | 5
  Not Hispanic or Latino | 25 | 17 | 42
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 22 | 13 | 35
  More than one race | 2 | 3 | 5
  Unknown or Not Reported | 1 | 0 | 1
ODSIS [Mean (Standard Deviation); unit: units on a scale] — Overall Depression Severity and Impairment Scale Total scores range from 0-20 with higher scores indicating more severe depression
  units on a scale | 8.90 (5.18) | 9.06 (4.84) | 8.96 (5.00)
PHQ-9 [Mean (Standard Deviation); unit: units on a scale] — Patient Health Questionnaire-9 Total score ranges from 0-27, with higher scores indicating more severe depression
  units on a scale | 12.69 (6.79) | 12.89 (9.28) | 12.77 (6.67)
GAD-7 [Mean (Standard Deviation); unit: units on a scale] — Generalized Anxiety Disorder-7 Total scores range from 0-21, with higher scores indicating more severe anxiety
  units on a scale | 10.52 (5.13) | 9.28 (5.85) | 10.04 (5.39)
OASIS [Mean (Standard Deviation); unit: units on a scale] — Overall Anxiety Severity and Impairment Scale Total scores range from 0-20, with higher scores indicating more severe anxiety
  units on a scale | 9.03 (4.19) | 9.11 (4.24) | 9.06 (4.16)
BSS [Mean (Standard Deviation); unit: units on a scale] — Beck Scale for Suicidal Ideation Total scores range from 0-38, with higher scores indicating more severe suicidal ideation
  units on a scale | 3.85 (6.11) | 3.23 (5.41) | 3.61 (5.80)
CSS [Mean (Standard Deviation); unit: units on a scale] — Commitment to Sobriety Scale Total scores range from 5-30, with higher scores indicating greater commitment to sobriety
  units on a scale | 15.24 (4.95) | 16.72 (5.26) | 15.81 (5.06)
Craving Scale [Mean (Standard Deviation); unit: units on a scale] — Craving Scale Total scores range from 0-27, with higher scores indicating more severe craving
  units on a scale | 17.48 (6.64) | 14.83 (7.96) | 16.47 (7.21)
Past 30-day PDA [Mean (Standard Deviation); unit: percentage of days abstinent] — Percent of last 30 days abstinent Scores range from 0-100%, with higher scores indicating more days abstinent
  percentage of days abstinent | 51.84 (34.44) | 61.30 (36.61) | 55.46 (35.20)
Past-month NSSI (SITBI) [Count of Participants; unit: Participants] — Count of participants with at least one day in which they engaged in NSSI over the past month (from Self-Injurious Thoughts and Behaviors Interview)
  Participants | 1 | 2 | 3
Past-month SI (SITBI) [Count of Participants; unit: Participants] — Count of participants with at least one day of suicidal ideation in the past month (from Self-Injurious Thoughts and Behaviors Interview)
  Participants | 10 | 5 | 15

OUTCOME MEASURES:

1. Primary Outcome: Acceptability of Adding UP Group Intervention to TAU
Description: Participants in the UP condition will complete the Client Satisfaction Questionnaire (CSQ-8) at post-treatment to assess acceptability of and satisfaction with the experimental intervention. Range of the scale is 8 (minimum) to 32 (maximum), with higher scores indicating greater levels of satisfaction with treatment received.
Time Frame: At the end of the 8-week treatment period
Population: 13 participants who attended at least 1 Unified Protocol session completed the CSQ-8.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Unified Protocol + Treatment As Usual
Number analyzed (Participants) | 13
units on a scale | 28.0 (4.6)

2. Primary Outcome: Feasibility of Adding UP Group Intervention to TAU
Description: Percentage of participants who dropout from treatment during the 8 week study period in the UP+TAU condition will be compared to the percentage of those who drop out from treatment in the TAU condition.
Time Frame: 8-week treatment period
Population: Total numbers randomized to each condition
Measure: Count of Participants; unit: Participants
Arm/Group | Unified Protocol + Treatment As Usual | Treatment As Usual Alone
Number analyzed (Participants) | 29 | 18
Participants | 13 | 6
Statistical Analysis 1: Comparison: Unified Protocol + Treatment As Usual vs Treatment As Usual Alone; Test type: Superiority; p = 0.63, Chi-squared, Corrected; df=1; Chi-squared statistic value = 0.23

3. Secondary Outcome: OASIS
Description: Overall Anxiety Severity and Impairment Scale (OASIS) administered at post-treatment. Total scores range from 0-20; higher scores indicate higher levels of anxiety.
Time Frame: At the end of the 8-week treatment period
Population: Participants who completed the OASIS at the post-treatment assessment (means at post-treatment reported below).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Unified Protocol + Treatment As Usual | Treatment As Usual Alone
Number analyzed (Participants) | 16 | 11
units on a scale | 5.44 (2.80) | 6.82 (3.43)
Statistical Analysis 1: Comparison: Unified Protocol + Treatment As Usual vs Treatment As Usual Alone; Linear mixed effects models with random intercepts (as best practice likelihood ratio tests dropping random slopes and intercepts indicated that only random intercepts should be retained) were used, with restricted maximum likelihood estimation (REML) for missing data. Analyses were intent-to-treat so included all randomized participants (n=29 in the UP+TAU group and n=18 in the TAU alone group), regardless of whether or not they completed the mid- or post-treatment assessments; Test type: Superiority; p = 0.29, Mixed Models Analysis — p-value is for the model parameter of the condition-by-time interaction term; Slope = 0.72 — The treatment condition effect was determined by the model parameter of the condition-by-time interaction term

4. Secondary Outcome: Depressive Symptoms Scale (ODSIS)
Description: Measured with the Overall Depression Severity and Impairment Scale (ODSIS) at post-treatment. Total scores range from 0-20; higher scores indicate higher levels of depressive symptoms.
Time Frame: At the end of the 8-week treatment period
Population: Participants who completed the post-treatment assessments (means reported below).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Unified Protocol + Treatment As Usual | Treatment As Usual Alone
Number analyzed (Participants) | 16 | 11
score on a scale | 6.06 (4.54) | 4.73 (3.93)
Statistical Analysis 1: Comparison: Unified Protocol + Treatment As Usual vs Treatment As Usual Alone; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = .50, Mixed Models Analysis — p-value is for the model parameter of the condition-by-time interaction term; Slope = -0.56 — The treatment condition effect was determined by the model parameter of the condition-by-time interaction term

5. Secondary Outcome: Suicidal Ideation
Description: Measured with the Beck Scale for Suicidal Ideation (BSI) at post-treatment. Total scores range from 0-38; higher scores indicate higher levels of suicidal ideation.
Time Frame: At the end of the 8-week treatment period
Population: Participants who completed the post-treatment assessment (means reported below).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Unified Protocol + Treatment As Usual | Treatment As Usual Alone
Number analyzed (Participants) | 16 | 11
score on a scale | 2.88 (4.56) | 1.09 (2.47)
Statistical Analysis 1: Comparison: Unified Protocol + Treatment As Usual vs Treatment As Usual Alone; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.45, Mixed Models Analysis — p-value is for the model parameter of the condition-by-time interaction term; Slope = -1.96 — The treatment condition effect was determined by the model parameter of the condition-by-time interaction term. BSI scores were binarized (0 and >=1) for this analysis due to the non-normal distribution of this outcome

6. Secondary Outcome: Number of Participants Who Reported Nonsuicidal Self-injury in the Past Month
Description: Measured with the Self-Injurious Thoughts and Behaviors Interview (SITBI) at post-treatment.
Time Frame: At the end of the 8-week treatment period
Measure: Count of Participants; unit: Participants
Arm/Group | Unified Protocol + Treatment As Usual | Treatment As Usual Alone
Number analyzed (Participants) | 16 | 11
Participants | 1 | 0

7. Secondary Outcome: Commitment to Sobriety
Description: Measured with the Commitment to Sobriety Scale (CSS) at post-treatment. Total scores range from 5-30; higher scores indicate higher levels of commitment to sobriety.
Time Frame: At the end of the 8-week treatment period
Population: Participants who completed the post-treatment assessment (means reported below).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Unified Protocol + Treatment As Usual | Treatment As Usual Alone
Number analyzed (Participants) | 16 | 11
score on a scale | 16.88 (5.55) | 17.27 (6.90)
Statistical Analysis 1: Comparison: Unified Protocol + Treatment As Usual vs Treatment As Usual Alone; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.76, Mixed Models Analysis — p-value is for the model parameter of the condition-by-time interaction term; Slope = -0.19 — The treatment condition effect was determined by the model parameter of the condition-by-time interaction term

8. Secondary Outcome: Substance Craving
Description: Measured with a three-item craving scale at post-treatment. Total scores range from 0-27; higher scores indicate higher levels of substance craving.
Time Frame: At the end of the 8-week treatment period
Population: Participants who completed the post-treatment assessment (means reported below).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Unified Protocol + Treatment As Usual | Treatment As Usual Alone
Number analyzed (Participants) | 16 | 11
score on a scale | 12.88 (7.03) | 8.45 (6.01)
Statistical Analysis 1: Comparison: Unified Protocol + Treatment As Usual vs Treatment As Usual Alone; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = .21, Mixed Models Analysis — p-value is for the model parameter of the condition-by-time interaction term; Slope = -1.07 — The treatment condition effect was determined by the model parameter of the condition-by-time interaction term. Due to the non-normal distribution of the Craving Scale, scores on this measure were binarized (< 15 and >= 15) for this analysis

9. Secondary Outcome: Percentage of Past 30 Days Abstinent From Substances
Description: Operationalized with the percentage days abstinent (PDA) in the past 30 days, measured via Timeline Follow Back (TLFB) at post-treatment.
Time Frame: At the end of the 8-week treatment period
Population: Participants who completed the post-treatment assessment (means presented below).
Measure: Mean (Standard Deviation); unit: percentage of past 30 days abstinent
Arm/Group | Unified Protocol + Treatment As Usual | Treatment As Usual Alone
Number analyzed (Participants) | 16 | 11
percentage of past 30 days abstinent | 72.29 (28.77) | 68.89 (21.41)
Statistical Analysis 1: Comparison: Unified Protocol + Treatment As Usual vs Treatment As Usual Alone; Due to the non-normal distribution of the PDA variable, this variable was treated as binary (<50% and >=50%) for mixed models; however, due to the small numbers of participants (< 5) in certain cells of treatment condition (UP versus TAU) by time point, we ran into issues with convergence of linear mixed models. Thus, here we report the results from an independent samples t-test of means (percentage of past 30 days abstinent) at post-treatment (UP versus TAU); Test type: Superiority; p = 0.77, t-test, 2 sided; t statistic = 0.29

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during the active study period (baseline to post-treatment assessment). Because the "waiting be be randomized" period (between baseline and date of randomization) varied across participants, the total study period lasted between 2 and 6 months.
Description: Adverse events were collected at the mid- and post-treatment assessments, which happened at 4 and 8 weeks, respectively, after the date of randomization, via systematic assessment. Non-systematic assessment was also used to collect information about adverse events by reviewing participants' electronic health records weekly during the study period.
Groups:
- Not Randomized: Participants in this arm were enrolled and completed the baseline visit but never randomized.
Arm/Group | Unified Protocol + Treatment As Usual | Treatment As Usual Alone | Not Randomized
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/18 | 0/9
Serious Adverse Events (participants affected / at risk) | 3/29 | 4/18 | 2/9
Other Adverse Events (participants affected / at risk) | 13/29 | 8/18 | 0/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Unified Protocol + Treatment As Usual (N=29) | Treatment As Usual Alone (N=18) | Not Randomized (N=9)
Relapse to substances (resulting in inpatient treatment) (Psychiatric disorders) | 2 (2) | 1 (1) | 0 (0)
Relapse to substances (resulting in emergency department visit)) (Psychiatric disorders) | 0 (0) | 1 (2) | 0 (0)
Active suicidal ideation with plan (resulting in inpatient treatment) (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Active suicidal ideation with plan (without inpatient treatment) (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Increase in psychotic symptoms (resulting in inpatient treatment) (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Pseudoseizure (resulting in emergency department visit) (General disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Unified Protocol + Treatment As Usual (N=29) | Treatment As Usual Alone (N=18) | Not Randomized (N=9)
Relapse to substances (without medical attention) (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Substance use resulting in emergency department visit (not hospitalized) (Psychiatric disorders) | 1 (2) | 0 (0) | 0 (0)
Non-fatal overdose (without seeking medical attention) (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Entered intensive outpatient program for substance use (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Increased suicidal ideation or urges to engage in nonsuicidal self-injury (Psychiatric disorders) | 2 (2) | 3 (4) | 0 (0)
Increased depressive symptoms (Psychiatric disorders) | 7 (7) | 3 (3) | 0 (0)
Increased anxiety-related symptoms (Psychiatric disorders) | 2 (2) | 3 (3) | 0 (0)
Cognitively impaired in context of increased anxiety/substance use (resulting in emergency departmen (Psychiatric disorders) | 1 (2) | 0 (0) | 0 (0)
Increased manic symptoms (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Increased restlessness (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Increased binge eating (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Increased stress (related to study group participation) (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Increased stress (not study-related) (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Adverse reaction to non-study medication (General disorders) | 0 (0) | 1 (1) | 0 (0)
Flu (General disorders) | 1 (1) | 0 (0) | 0 (0)
Headaches/migraine (General disorders) | 1 (1) | 1 (1) | 0 (0)
Weight gain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Chest tightness attributed to onset of electronic cigarette use (General disorders) | 1 (1) | 0 (0) | 0 (0)
Head injury (General disorders) | 1 (1) | 0 (0) | 0 (0)
Contracted STD (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sleep apnea symptoms (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0)
Asthma symptoms (General disorders) | 0 (0) | 1 (2) | 0 (0)
Abdominal pain/nausea/vomiting (in context of early withdrawal) (General disorders) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Due to dropout, there were small numbers of participants analyzed at post-treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-09-18): https://cdn.clinicaltrials.gov/large-docs/08/NCT03315208/SAP_000.pdf
  • Study Protocol (2019-07-05): https://cdn.clinicaltrials.gov/large-docs/08/NCT03315208/Prot_001.pdf